CLINICAL TRIAL: NCT05575102
Title: Walking Football for People With Chronic Breathlessness: a Mixed-methods Feasibility Study
Brief Title: Walking Football for People With Chronic Breathlessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Samantha Harrison, Professor of Respiratory Rehabilitation, Teesside University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10814
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Dyspnea
Keywords: Dyspnea; Chronic Breathlessness; Football; Walking; Exercise; Physical Activity; Pulmonary Rehabilitation; Feasibility; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Dyspnea; Motor Activity; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking Football (Experimental): Walking football intervention for 6-weeks (2-hour per week) at a local sports hall, supervised by a walking football coach with assistance from CB.
  Interventions: Other: Walking Football

INTERVENTIONS:
Other: Walking Football — Walking Football (Soccer): Typical football rules apply but without running.
  Participants will play at a local sports hall for 6-weeks, (2-hour per week). Time will be split between warm-up, football practice drills, and small-sided games.

SUMMARY:
The objective of this study is to evaluate the feasibility of a walking football intervention for people with chronic breathlessness. Chronic breathlessness refers to breathlessness that persists despite optimal treatment of the underlying pathophysiology. Roughly 9-13% of the general population will experience chronic breathlessness, with incidence rising with age to 37% for those aged over 60years.

This mixed-methods study will offer patients who have enrolled on to pulmonary rehabilitation (PR) the prospect to partake in walking football once they have completed their scheduled programmes (or voluntarily dropped-out); introducing a potential opportunity for long-term exercise maintenance post PR. Participants will be recruited from North Tees & Hartlepool Foundation Trust, and South Tees Foundation Trust.

PR is recommended for all people with chronic breathlessness and has been shown to improve exercise capacity and health-related quality of life. However, PR programmes typically only last for 6-12 weeks, and have little to no impact on long-term physical activity levels. Walking Football has been identified as a potential form of exercise which people with breathlessness could maintain post-PR, thus offering a solution to PRs limited ability to promote exercise maintenance.

Participants will be invited to play walking football for 6-weeks (2-hours weekly) in the Middlesbrough/Stockton area. Before and after weeks 1 and 6, breathlessness-relevant outcomes will be measured including; exercise capacity, lower-limb strength, perceived breathlessness, quality of life, balance confidence, depression, and anxiety.

During a participant's third session, one-time physical intensity outcomes will be calculated during play including heart-rate and perceived intensity. Participants will also be invited to an interview to discuss how feasible they have found the football, any benefits they may have experienced, and how the football programme could be improved.

The study will officially end with a co-production workshop; a focus group with stakeholders (players, physiotherapists, co-ordinators, researchers) after preliminary analysis has been conducted to discuss initial findings.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of chronic breathlessness via a chronic respiratory condition (through referral to PR)

  * Example conditions include; COPD, severe asthma, Pulmonary Fibrosis, Lung Disease (This does not include Long Covid as many patients often make a full recovery over time).
* Be 35 years or over at the point of recruitment
* Scheduled PR programme ends within the recruitment window
* Be able to communicate with good verbal English or use adaptive equipment to communicate
* Respiratory condition is stable (e.g. six weeks clear of exacerbation in COPD)

Exclusion Criteria:

* Unstable Angina
* Other conditions that may affect balance (e.g. neurological)
* Recent exacerbation of COPD (within the last six weeks)
* Unable to provide written informed consent
* Unable to speak English or no translation options available
* Any other acute health conditions that would make activity unsafe e.g. acute infection

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Recruitment and Consent Rate | 6-Months
  Percentage of eligible participants given an information sheet who consent to participate
Completion Rate | 6-Weeks
  Percentage of participants who complete at least four of the available six sessions
Methodology and Intervention Acceptability | 10-Weeks
  Percentage of participants who complete all pre-post outcome measurements, intensity outcome measurements, and partake in an interview.
Adverse Events | 6-Weeks
  Number of Serious and Minor Adverse Events recorded

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Harrison, Principal Investigator — Teesside University
Locations (1):
- Tesside University, Middlesbrough, United Kingdom